CLINICAL TRIAL: NCT02348294
Title: Measurement of Cytokines, Bloodflow and Erythema Index After Pressure and Shear- Force Loading in Patients With Diabetes Mellitus Type 2
Brief Title: The Effect of Shear- Force at the Skin in Patients With Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: NL50794.068.14
Record Dates: First submitted 2015-01-22; First posted 2015-01-28 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Pressure Ulcer; Diabetes Mellitus Type 2; Charcot- Osteoarthropathy
MeSH Terms: conditions — Pressure Ulcer; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Healthy volunteers (Other): Shear- force 19 newton and 3,9 kpa pressure for half an hour
  Interventions: Other: Shear- force 19 newton and 3,9 kpa pressure for half an hour
- Diabetes Mellitus type 2 without neuropathy (Other): Shear- force 19 newton and 3,9 kpa pressure for half an hour
  Interventions: Other: Shear- force 19 newton and 3,9 kpa pressure for half an hour
- Diabetes Mellitus type 2 with neuropathy (Other): Shear- force 19 newton and 3,9 kpa pressure for half an hour
  Interventions: Other: Shear- force 19 newton and 3,9 kpa pressure for half an hour
- Charcot Osteoarhtopathy (Other): Shear- force 19 newton and 3,9 kpa pressure for half an hour
  Interventions: Other: Shear- force 19 newton and 3,9 kpa pressure for half an hour

INTERVENTIONS:
Other: Shear- force 19 newton and 3,9 kpa pressure for half an hour

SUMMARY:
1. The objective of this study is to acquire knowledge about the development of reactive hyperaemia and inflammatory responses of the skin after shear- force and pressure loading. We want to investigate if patients with diabetes type 2 will develop more skin damage, because of a decreased microvascular function.
2. The second objective of this study is: to investigate if the cytokine production of the skin is increased in patients with type 2 diabetes with a history of Charcot osteoarthropathy in comparison with patients with neuropathy without a history of Charcot osteoarthropathy.

The participant is asked to put his left arm on a support cushion. Then we mark an area of 2.5 cm x 3 cm with a permanent marker at the plantar aspect of the left fore-arm and the adhesive side of a Sebutape is placed within this area for collection of IL-1α/ total protein concentrations in a non- loaded situation (event 1) for two minutes. Second, we measure the cutaneous blood cell flux within the borders of the marked area with a Laser doppler. Finally, we measure the erythema index in this area with a colorimeter. Then we place the shear- pad over the marked area we apply 9,8 Newton (N) pressure with 19 N shear- force for half an hour. After this period a new Sebutape is placed for two minutes, followed by cutaneous blood cell flux and the erythema index measurement within the borders of the marked area. We repeat these measures after 15 minutes, 30 minutes, 45 minutes and 60 minutes, At the same time we performed the same experiment at the right arm, but instead of loading this arm with shear- force and pressure, we apply only 9,8 N pressure at this arm. The same measures with the sebutape, laser doppler and colorimeter are done before and after loading of the skin. The measures are repeated at 15 minutes, 30 minutes, 45 minutes and 60 minutes.

DETAILED DESCRIPTION:
1. Pressure ulcers, also known as bedsores occurs as a result of mechanical loading (combination of pressure and shear- force) of the skin. We proved that IL-1alpha (measurement of skin damage) and reactive hyperaemia (RH) are increased after a combined loading of pressure and shear- force with our own developed shear- force model. This RH is probably a protective mechanism of the loaded skin and is clinically seen as blanchable erythema. Blanchable erythema is seen as an important risk indicator for the development of pressure ulcers. Patients with Diabetes Mellitus type 2, however, will develop less blanchable erythema (RH), because of a decreased micro vascular function. Therefore, they will get less preventive measures against pressure ulcers. We do expect, however, that more skin damage occurs when RH is decreased, so we want to investigate if patients with type 2 diabetes (with or without neuropathy) will develop less RH and more skin damage (IL-1alpha) after shear force application at the skin compared with healthy volunteers.
2. Charcot- neuro- osteoarthropathy is a rare, but serious complication of polyneuropathy. Most of the times it occurs at the feet in patients with diabetes with neuropathy. It is associated with inflammation, hyperaemia, bone deformation and luxation of the joints. The pathogenesis is not well understood: the hyperemic response of the skin to external stimuli is increased, but we do not know if this hyperaemia is a result of primary hypervascularity or a increase in primary cytokines. Our research model gives us the opportunity to investigate if: the local cytokine production is increased in patients with diabetes type with neuropathy and a history of charcot osteoarthropathy after shear- force application at the skin compared with patients with type 2 diabetes with neuropathy.

Study population:

Group A:

* Healthy volunteers
* > 40 years

Group B;

* patients with Diabetes Mellitus type 2 (DM) without neuropathy
* age > 40 years
* Valk score < 4

Group C:

* Patients with DM type 2 with neuropathy
* age > 40 years
* Valk score > 4

Group D

* Patients with (pre)- existing Charcot Osteoarhtropathy
* age > 40 years
* Valk score > 4 Primary study parameters/outcome of the study

  1. IL-1 α/ total protein ratio
  2. Bloodflow of the skin (in flux )
  3. Erythema index of the skin

The participant is asked to put his left arm on a support cushion. Then we mark an area of 2.5 cm x 3 cm with a permanent marker at the plantar aspect of the left fore-arm and the adhesive side of a Sebutape is placed within this area for collection of IL-1α/ total protein concentrations in a non- loaded situation (event 1) for two minutes. Second, we measure the cutaneous blood cell flux within the borders of the marked area with a Laser doppler. Finally, we measure the erythema index in this area with a colorimeter. Then we place the shear- pad over the marked area we apply 9,8 Newton (N) pressure with 19 N shear- force for half an hour. After this period a new Sebutape is placed for two minutes, followed by cutaneous blood cell flux and the erythema index measurement within the borders of the marked area. We repeat these measures after 15 minutes, 30 minutes, 45 minutes and 60 minutes, At the same time we performed the same experiment at the right arm, but instead of loading this arm with shear- force and pressure, we apply only 9,8 N pressure at this arm. The same measures with the sebutape, laser doppler and colorimeter are done before and after loading of the skin. The measures are repeated at 15 minutes, 30 minutes, 45 minutes and 60 minutes.

Outcomes; IL-1alpha/ total protein- ratio Cutaneous blood cell flux Erythema index

ELIGIBILITY:
Inclusion Criteria:

* Group A:
* Healthy volunteers
* > 40 years

Group B;

* patients with Diabetes Mellitus type 2 (DM) without neuropathy
* age > 40 years
* Valk score < 4

Group C:

* Patients with DM type 2 with neuropathy
* age > 40 years
* Valk score > 4

Group D

* Patients with (pre)- existing Charcot Osteoarhtropathy
* age > 40 years
* Valk score > 4

Exclusion Criteria:

* Trauma fore arms
* Skin diseases (psoriasis, eczema)
* NSAID use in last seven days
* Bèta blocker use
* Corticosteroids
* Auto- immune diseases
* Muscular dystrophy
* Malignancy
* Participant is unable to give informed consent
* Peripheral artery disease (doppler eai <0.9)
* Hab1c percentage last 3 months > 11%

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Increase in IL-1alpha/ total protein ratio | 0, 15, 30, 45, 60 minutes after intervention
Increase in Cutaneous blood cell flux | 0, 15, 30, 45, 60 minutes after intervention
Increase in erythema index | 0, 15, 30, 45, 60 minutes after intervention